CLINICAL TRIAL: NCT03920813
Title: Determinants of Mercaptopurine Toxicity in Paediatric Acute Lymphoblastic
Brief Title: Determinants of Mercaptopurine Toxicity in Paediatric Acute Lymphoblastic Leukemia Maintenance Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018Mercaptopurine001
Record Dates: First submitted 2019-04-15; First posted 2019-04-19 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Antitumor drugs (Experimental): Mercaptopurine administered at standard dose for children with hematological neoplasms.
  Interventions: Drug: Mercaptopurine

INTERVENTIONS:
Drug: Mercaptopurine — Dose of mercaptopurine was adjusted to maintain a target white blood cells (WBC) between 2.0-3.0 × 109/L.
  Other Names: Purinethol

SUMMARY:
The present study was conducted to assess the population pharmacokinetics of 6-mercaptopurine (6-MP) in Pediatric Acute Lymphoblastic Leukemia (ALL) and genetic polymorphisms

DETAILED DESCRIPTION:
The investigators' purpose was to identify genetic factors and metabolite concentrations associated with both hematological toxicity in patients with ALL maintained on 6-MP in Chinese.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been diagnosed with Acute Lymphoblastic Leukemia
* Childhood patients who were undergoing chemotherapy or continuous follow-up after completion of chemotherapy
* Patients received the phase of maintenance therapy that included oral 6-MP (>4 weeks) and completion of ≥ 6 months according to the CCLG (Chinese Children's Leukemia Group) protocol-ALL 2015

Exclusion Criteria:

* Patients with high-risk ALL (presence of higher-risk features: MRD ≥ 1% at 46 day, or age < 6 month and white blood cell (WBC) count ≥ 300×109/L with translocations t(9;22) (q34;q11) [BCR-ABL], t(4;11) (q21;q23) [AF4/MLL], t(1;19) (q23;p13) [E2A-PBX1] or other MLL-rearrangements) were removed

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Red blood cells (RBC) concentration of 6-mercaptopurine (6-MP) | at second day after oral administration
  To detect of RBC 6-MP metabolite concentrations and evaluate the association of metabolite concentrations and side effects
Genetic polymorphisms in Chinese patients with ALL | at second day after oral administration
  To detect the frequencies of genetic polymorphisms of Chinese patients receiving 6-MP for treatment of ALL

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Principal Investigator — Shandong University